CLINICAL TRIAL: NCT04090034
Title: Peptide Receptor Radionuclide Therapy (PRRT) for the Treatment of Neuroendocrine
Brief Title: Peptide Receptor Radionuclide Therapy (PRRT) for the Treatment of Neuroendocrine Tumors
Acronym: PRRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 022.HPB.2019.D
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-03

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treated w PRRT: Patients who received treatment of gastroenteropancreatic primary NETs with PRRT per the treating physicians discretion.
  Interventions: Procedure: Peptide Receptor Radionuclide Therapy

INTERVENTIONS:
Procedure: Peptide Receptor Radionuclide Therapy — a molecular therapy (also called radioisotope therapy) used to treat a specific type of cancer called neuroendocrine tumors or NETs

SUMMARY:
The specific aim is of this study is to gain a better understanding of the patient characteristics, treatment responses, survival outcomes, and adverse events associated with PRRT in patients with gastroenteropancreatic primary NETs.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) make up a large range of malignancies that arise from neuroendocrine cells in multiple organs of the body. Hallet et al conducted a large population-based study that demonstrated that 21% of NET patients presented with metastatic disease and another 38% developed metastases after resection of the primary tumor (Hallet et al., 2015). This burden demonstrates the need for effective systemic therapy for advanced NETs. Options for systemic therapy include peptide receptor radionuclide therapy (PRRT).

A need for more prospective series are needed on treatment responses and survival outcomes related to gastroenteropancreatic primary NETs treated with PRRT was identified. Thus the purpose of this study is to collect clinical data related to treatment of gastroenteropancreatic primary NETs s with PRRT. Clinical data related to patient characteristics, treatment responses and survival outcomes related to the treatment of gastroenteropancreatic primary NETs with PRRT and on adverse events and complications related to PRRT treatment will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Diagnosed with gastroenteropancreatic primary NET and has consented to undergo PRRT per the treating physician. Specifically:

   * Will consider other primaries on a case by case basis if dotatate scan (+) and meet all other criteria.
   * Metastatic or Locally Advanced AND Inoperable
   * Clear disease progression on Octreotide over less than 3 years (RECIST 1.1)
   * Presence of disease within 24 weeks as identified by PET/CT scans with Ga-68 DOTATATE reporting the Krenning score for low-grade NET and/or PET/CT scans with FDG for transformation to high-grade NET
   * Well differentiated on path - Ki67 < 20%
   * Octreotide positive on pathology (if not documented, acceptable if PET/CT imaging shows lesions with Ga-68 DOTATATE uptakeLabs:

     * Cr. <1.7
     * Hgb >8
     * WBC >2K
     * Plt >75K
     * Bili < 3x normal limit
   * No Octreotide within 30 days of administration.
3. Willing and able to comply with the protocol requirements
4. Able to comprehend and sign the Informed Consent Form in English.

Exclusion Criteria:

* Do not meet the Study Inclusion Criteria laid out in section 6.3

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be screened for NETs per standard of care. Those patients, who have or will undergo the PRRT procedure, will be offered the opportunity to participate in this registry study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-28 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Demographics and other patient data | 7 years from date of procedure
  (such as age at diagnosis, sex, history of smoking alcohol use and symptoms at the time of diagnosis)
Tumor specific data | 7 years from date of procedure
  Tumor site, tumor grade, stage, presence of tumor necrosis, number of mitoses and percentage of Ki-67 and MIB-1 positive cells (proliferative index)
Use of somatostatin analogs | 7 years from date of procedure
  at the time of PRRT, location, isotope used and dose of isotope for each PRRT
Biomarker data (chromogranin A and pancreastatin) | 7 years from date of procedure
  at the time of diagnosis, before and after the first PRRT, and after the second PRRT were also extracted
Diagnostic imaging findings | 7 years from date of procedure
  prior to PRRT and response after PRRT, date of progression on imaging after PRRT, and status of disease on imaging at the last follow-up were also recorded
Overall survival (OS) | 7 years from date of procedure
  the time from diagnosis to death of any cause.
Time to progression (TTP) | 7 years from date of procedure
  the time from the first PRRT until any progression on diagnostic imaging
Treatment responses and progression | 7 years from date of procedure
  assessed with cross-sectional imaging with either computerized tomography (CT) or magnetic resonance imaging (MRI) or positron emission tomography (PET) or single-photon emission computed tomography (SPECT).
Response | 7 years from date of procedure
  any response of any magnitude
Disease progression | 7 years from date of procedure
  any increase in lesion sizes and/or appearance of new metastatic lesions on diagnostic imaging exams.
Adverse events | 7 years from date of procedure
  will be assessed by the investigator who will determine whether or not the event is related to PRRT or related to progression of disease (gastroenteropancreatic primary NET), and whether or not the event meets serious criteria. AEs related to PRRT will be recorded in the study registry.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Mejia, MD, Principal Investigator — Liver Institute at Methodist Dallas Medical Center
Locations (2):
- United States (2):
  - Clinical Research Institute at Methodist Health System, Dallas, Texas
  - Methodist Dallas Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided